CLINICAL TRIAL: NCT01643863
Title: A Multi-center Non-interventional Study in Rheumatoid Arthritis (RA) Patients Treated With Tocilizumab (TCZ)
Brief Title: A Non-Interventional Study of RoActemra/Actemra (Tocilizumab) in Monotherapy in Patients With Rheumatoid Arthritis (MONACO)
Status: Terminated | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML28202
Record Dates: First submitted 2012-07-16; First posted 2012-07-18 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cohort

SUMMARY:
This multi-center observational study will evaluate the use of RoActemra/Actemra (tocilizumab) in monotherapy in patients with rheumatoid arthritis. Eligible patients initiated on RoActemra/Actemra treatment according to the licensed label will be followed for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/= 18 years of age
* Moderate to severe rheumatoid arthritis according to the revised (1987) ACR criteria
* Patients in whom the treating physician has made the decision to commence RoActemra/Actemra treatment in monotherapy, in case of methotrexate intolerance or when continuous methotrexate treatment is inadequate (in accordance with the local label), and who have received (or started) RoActemra/Actemra monotherapy treatment within 8 weeks prior to the enrolment visit.
* Concomitant corticosteroids (oral or intra-articular) or non-steroidal anti-inflammatory drugs (NSAIDs) are allowed

Exclusion Criteria:

* Patients in whom RoActemra/Actemra is contraindicated according to the approved Summary of Product Characteristics
* Patients who have received RoActemra/Actemra more than 8 weeks prior to the enrolment visit
* Patients who have previously received RoActemra/Actemra in a clinical trial or for compassionate use
* Concomitant DMARD treatment for rheumatoid arthritis (e.g. hydroxychloroquine, sulfasalazine, methotrexate, leflunomide, gold compounds, cyclosporine) when starting treatment with RoActemra/Actemra
* Treatment with any investigational agent within 4 weeks (or 5 half-lives of the investigational agent, whichever is longer) before starting treatment with RoActemra/Actemra
* History of autoimmune disease or any joint inflammatory disease other than rheumatoid arthritis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with rheumatoid arthritis initiated on treatment with RoActemra/Actemra in monotherapy
Sampling Method: Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2012-08; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Proportion of patients on RoActemra/Actemra at 6 months | approximately 20 months

SECONDARY OUTCOMES:
Rates of dose modifications/interruptions | approximately 20 months
Clinical/demographic patient characteristics at initiation of RoActemra/Actemra treatment | approximately 20 months
Efficacy: Response according to total joint count evaluation by DAS28/EULAR/SDAI/CDAI/ACR | approximately 20 months
Physician Global Assessment of disease activity | approximately 20 months
Patient reported outcomes: Health Assessment Questionnaires | approximately 20 months
Introduction/use of disease-modifying anti-rheumatic drugs (DMARDs) | approximately 20 months
Time to reduction/withdrawal of corticosteroids | approximately 20 months
Safety: Incidence of adverse events\n | approximately 20 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (2):
- Portugal (2):
  - Lisbon
  - Porto